CLINICAL TRIAL: NCT00198809
Title: Use of Herbal Supplements in Weight Loss and Weight Maintenance
Status: Terminated | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Wellness International, Ltd. (Unknown)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: WELL2001-01
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2005-09-20 (Estimated); Status verified 2004-04

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — Nutrition Assessment

INTERVENTIONS:
Drug: Biolean + Diet education
Drug: Biolean Free + Diet education
Drug: Placebo + Diet education

SUMMARY:
Effects of herbal products on weight loss, weight maintenance and metabolic rate.

* The objective of this study is to evaluate the efficacy of two herbal weight loss products, BioLean and BioLean Free compared to each other and a matching placebo, in effects on appetite suppression, changes in metabolism, weight loss, and safety in overweight men and women over a 12 month active weight loss and weight maintenance program.
* This is a randomized double-blind study. The planned sample size is 180 healthy, overweight (BMI 27-40) males and females aged 18-60.

DETAILED DESCRIPTION:
• The study data collection will occur in two phases, active weight loss (phase 1) and weight maintenance (phase 2). Transition into phase 2 will be individually determined by participant attainment of a goal 'healthy' weight. During the 52 weeks participants will pick up supplemental pills, have weight measured, and meet for educational meeting on an every other week basis. Upon entering phase 2, participants will have the option of educational sessions on a monthly basis or every other week. Participants will have a goal 'healthy' weight determined at baseline by a combination of personal goals, Harris Benedict Equation goals, body composition goals, and BMI range. All participants will be put on a weight reduction plan to reach these goals and be randomly assigned to one of 3 treatment groups, Biolean, Biolean Free, or Placebo. Since it is expected some participants will reach goal weight before others, the 2nd milestone data collection will occur at attainment of goal weight. To assure all participants have 3 data collection points, any participant who is not expected to reasonably reach their goal weight by 34 weeks will have the 2nd milestone data collection at 26 weeks. The 3rd milestone data collection for all participants is 52 weeks after initial intake of supplement. Upon attainment of goal weight and 2nd data collection point, participants will be educated on a weight maintenance plan and given a new meal plan to achieve long term healthy weight maintenance.

ELIGIBILITY:
Inclusion Criteria:

Between 18-60 years of age, overweight (Body Mass Index between 27-40) and desiring weight loss, normal EKG (electrocardiogram), not using or on a stable dosage of appetite- affecting medications (e.g., Prozac or other SSRIs, Synthroid, steroids), non-pregnant at screening by serum pregnancy test if female of childbearing capacity and using an acceptable method of birth control (tubal ligation, abstinence, properly used condom or diaphragm, oral or implanted contraceptives, or intrauterine device) To be considered not childbearing potential, participant must be at least one year post-menopausal or surgically sterile, willing and able to comply with the protocol requirements, willing and able to give informed consent, have a regular source of health care and permission of primary care provider.

Exclusion Criteria:

Chronic health problems (not including obesity, allergies, skin problems, or occasional GERD or IBS symptoms). Participant may not have bulimia or laxative abuse, substance abuse, or alcohol intake > 10 oz. per week, or be under treatment for a psychiatric disorder (including depression, bipolar disorder, and anxiety determined by self-report during phone screening and the Beck Inventory survey to be completed during screening visit), as determined at screening. Use of ephedrine-containing products in the past 3 months, unwillingness to limit use of caffeinated beverages to three cups per day during participation in the study, active cigarette smoking of > 1 cigarette per week, resting systolic blood pressure > 140 mmHg or diastolic > 90 mmHg or pulse < 55 or > 100, and if female pregnant or breast-feeding.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 250
Dates: Start 2002-11; Study Completion 2004-02

PRIMARY OUTCOMES:
weight
blood pressure
pulse
blood

SECONDARY OUTCOMES:
psychometrics
body composition

CONTACTS AND LOCATIONS:
Overall Officials: Lawrence J Cheskin, MD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (1):
- Johns Hopkins Bloomberg School of Public Health, Baltimore, Maryland, United States